CLINICAL TRIAL: NCT05809960
Title: The Effect of Nursing Support Program Developed in Accordance With Roy Adaptation Model for Women in Surgical Menopause on Their Life Quality
Brief Title: The Effect of Nursing Support Program for Women in Surgical Menopause on Their Life Quality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mehtap Gümüşay (Other)
Responsible Party: Sponsor-Investigator, Mehtap Gümüşay, Principal Investigator, Ordu University
Organization: Ordu University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: OrduU-SBF-MG-1
Record Dates: First submitted 2023-03-30; First posted 2023-04-12 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-03

CONDITIONS: Nursing Caries; Surgical Menopause; Quality of Life
Keywords: Nursing support program; Roy Adaptation Model; Depressive symptom status; Sleep quality
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Investigation Group (Experimental): Education was given, which was prepared in line with the Roy Adaptation Theory and considering the literature, including the problems experienced in menopausal periods and the approaches used to cope with them. The progressive relaxation exercise was explained and taught to the women and the first application was provided with the instructions. "Menopause and Life" booklet prepared in line with Roy Adaptation Theory was given to support the education given and to remember the information afterwards.
  Interventions: Other: Nursing support program
- Control Group (Active Comparator): Routine nursing care was given to the control group. The clinical routine has not been exceeded.
  Interventions: Other: Routine nursing care

INTERVENTIONS:
Other: Nursing support program — It was discussed about the operation and surgical menopause that the woman will undergo after hospitalization for the operation. Education was given including the problems experienced during menopause and the approaches used to cope with them. Progressive relaxation exercises were taught and practiced. In order to carry out these procedures, an interview of approximately 45-60 minutes was held with each woman. During the program, four planned meetings were held. One of them was face-to-face and the others were phone calls. During the phone calls, the symptoms experienced by the women and their coping methods were discussed and the questions of the women were answered. The average of each phone call was 20-30 minutes.
  Arms: Investigation Group
Other: Routine nursing care — Routine nursing care was given to the control group. The clinical routine has not been exceeded. It includes discharge training for the surgery.
  Arms: Control Group

SUMMARY:
Objective: The aim of this study was to determine the effect of the nursing support program developed in line with the Roy Adaptation Model on the quality of life, sleep quality and depressive symptom status of women in surgical menopause.

Design: The study was a single-center, randomized, controlled trial. Setting: This study was carried out in the gynecology clinic of a training and research hospital in Türkiye.

Method: The participants were randomized into two equal groups: intervention and control. The nursing support program developed in addition to routine nursing care was applied to the intervention group. Routine nursing care was given to the women in the control group. Data were collected with "Personal Information Form", "Menopause-Specific Quality of Life Questionnare", "Pittsburgh Sleep Quality Index" and "Perimenopausal Depression Scale".

Hypothesis:

H0-a: Nursing support program developed in line with the Roy Adaptation Model has no effect on the quality of life of women who have undergone surgical menopause.

H0-b: Nursing support program developed in line with the Roy Adaptation Model has no effect on the sleep quality of women who have undergone surgical menopause.

H0-c: Nursing support program developed in line with the Roy Adaptation Model has no effect on the depressive symptom status of women who have undergone surgical menopause.

ELIGIBILITY:
Inclusion Criteria:

* To have undergone surgical menopause
* To be literate
* To agree to participate in the study

Exclusion Criteria:

* To have natural menopause before the operation
* To have an oncological disease
* To have a psychiatric disease
* To use sleeping pills
* To use hormonal therapy
* To have physical and mental disability
* To have barrier to communication

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 77 (Actual)
Dates: Start 2020-01-20 (Actual); Primary Completion 2021-02-18 (Actual); Study Completion 2021-07-30 (Actual)

PRIMARY OUTCOMES:
Life quality | 6 months
  Women's quality of life was evaluated with the Menopause-Specific Quality of Life Questionnaire. The questionnaire consists of 4 sub-dimensions. The score for each dimension is calculated separately. High scores from the questionnaire indicate low quality of life.
Sleep quality | 6 months
  Sleep quality of women was evaluated with the Pittsburgh Sleep Quality Index. The index consists of 7 sub-dimensions. The score for each dimension is calculated separately.
Depressive symptom status | 6 months
  Depressive symptom status of women was evaluated with the Perimenopausal Depression Scale. The scale consists of 5 subscales. Minimum point is "0" an maximum point is "48".

CONTACTS AND LOCATIONS:
Locations (1):
- Ordu University, Ordu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No